CLINICAL TRIAL: NCT05634590
Title: The Efficacy and Safety of Fruquintinib Combined With FOLFIRI/FOLFOX as Second-line Treatment in Patients With RAS-mutant Metastatic Colorectal Cancer: A Single-center, Open-label, Single-arm Study
Brief Title: The Efficacy and Safety of Fruquintinib Plus FOLFIRI/FOLFOX as Second-line Treatment in Patients With RAS-mutant Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Xu, Professor, Chief of Department of Colorectal Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C119
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Fruquintinib plus Chemotherapy; RAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; IFL protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib plus FOLFIRI/FOLFOX (Experimental): Patients will receive fruquintinib plus FOLFIRI/FOLFOX. Oxaliplatin-based or irinotecan-based chemotherapy depending on previous chemotherapy (chemotherapy switch).
  Interventions: Drug: Fruquintinib; Drug: FOLFIRI; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Fruquintinib — 4mg, orally, once daily, 3 weeks on/ 1 week off
Drug: FOLFIRI — Irinotecan 180 mg/m2, and LV 400 mg/m2 followed by bolus 5-fluorouracil 400mg/m2 and a 46-48h continuous infusion 2400mg/m2 5-fluorouracil on day 1, q2w
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m2, and LV 400 mg/m2 followed by bolus 5-fluorouracil 400mg/m2 and a 46-48h continuous infusion 2400mg/m2 5-fluorouracil on day 1, q2w

SUMMARY:
RAS mutations are found in nearly half of colorectal cancer patients. However, there is no targeted driver gene drugs have been approved for RAS-mutated patients. For RAS mutant metastatic colorectal cancer, the commonly used treatment regimen is bevacizumab combined with chemotherapy.

DETAILED DESCRIPTION:
This is a single-center, open, single-arm study exploring the efficacy and safety of fruquintinib combined with FOLFIRI/FOLFOX in the treatment of RAS-mutated metastatic colorectal cancer (mCRC) who failed standard therapy. Patients will receive fruquinitinib combined with chemotherapy (FOLFOX or FOLFIRI regimens), which depend on the previous chemotherapy regimen (chemotherapy switch).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Histological or cytological confirmed colorectal cancer;
* RAS mutation
* Expected survival >12 weeks;
* Fail in previous standard therapy, which must include FOLFOX/FOLFIRI;
* ECOG PS 0-1;
* At least one measurable lesion (according to RECIST1.1);
* Adequate hepatic, renal, heart, and hematologic functions;
* Negative serum pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

* Received other investigational drugs within 4 weeks prior to treatment;
* Prior treatment with anti-angiogenic small molecule targeted drugs, such as fruquintinib, etc;
* Symptomatic brain or meningeal metastases (except for patients with BMS who have received local radiotherapy or surgery for more than 6 months and whose disease is stable);
* Severe infection (e.g., requiring intravenous antibiotics, antifungal drugs, or antiviral drugs) within 4 weeks prior to treatment;
* Patients with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
* Patients who had active bleeding or coagulopathy within 2 months before enrollment, had a tendency to bleed, or were receiving thrombolytic therapy and were considered by the investigator to be ineligible for enrollment;
* Active heart disease, including myocardial infarction, severe/unstable angina, 6 months prior to treatment. Echocardiography examination left ventricular ejection fraction < 50%, arrhythmia control is not good;
* The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Allergy to the study drug or any of its excipients;
* The patient is unable to take the drug orally, or the patient has a condition judged by the investigator to affect the absorption of the drug;
* Women who are pregnant (with a positive pregnancy test before medication) or breastfeeding;
* Urine routine showed urine protein ≥2+, and 24-hour urine protein level >1.0g;
* Other conditions deemed by the investigator to be ineligible for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | assessed up to 1 year
  time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
Objective response rate (ORR) | assessed up to 1 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.
Disease Control Rate (DCR) | assessed up to 1 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Overall survival (OS) | assessed up to 2 year
  time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Caner Center, Shanghai, Shanghai Municipality, China